CLINICAL TRIAL: NCT03981094
Title: An Open Label Study to Assess the Pharmacokinetic Interaction Between Pirfenidone and BMS-986278 Following a Single Oral Dose Administration in Healthy Participants
Brief Title: A Study of the Pharmacokinetic Interaction Between Pirfenidone and BMS-986278 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IM027-041
Record Dates: First submitted 2019-05-21; First posted 2019-06-10 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — pirfenidone

STUDY DESIGN:
Intervention Model Description: The study will be conducted in three periods, so that all the randomized participants receive treatment (participants receive pirfenidone only, or BMS-986278 only, or both together during each treatment period).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BMS-986278 (Experimental)
  Interventions: Drug: BMS-986278
- Pirfenidone (Experimental)
  Interventions: Drug: Pirfenidone
- BMS-986278 + Pirfenidone (Experimental)
  Interventions: Drug: BMS-986278; Drug: Pirfenidone

INTERVENTIONS:
Drug: BMS-986278 — suspension
  Arms: BMS-986278; BMS-986278 + Pirfenidone
Drug: Pirfenidone — capsule
  Arms: BMS-986278 + Pirfenidone; Pirfenidone

SUMMARY:
The main objectives of this study are to characterize the PK of BMS-986278 after administration of a single dose of BMS-986278 alone or in combination with pirfenidone, as well as to characterize the PK of pirfenidone after administration of a single dose of pirfenidone alone or in combination with BMS-986278

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent.
* Healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.

Exclusion Criteria:

* Women of child bearing potentia (WOCBP), pregnant or breastfeeding.
* History of significant cardiovascular disease.
* Participants who have smoked or used smoking cessation or nicotine containing products within 3 months of the first dose of study.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed serum concentration (Cmax) of BMS-986278 and pirfenidone alone or in combination | Up to day 5 of each period (Each period is 7 days; 3 periods total)
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration [AUC(0-T)] of BMS-986278 and pirfenidone alone or in combinaton | Up to day 5 of each period (Each period is 7 days; 3 periods total)
Area under the plasma concentration-time curve extrapolated to infinity [(AUC(INF)] of BMS-986278 and pirfenidone alone or in combinaton | Up to day 5 of each period (Each period is 7 days; 3 periods total)

SECONDARY OUTCOMES:
Incidence of AEs (adverse events), SAEs (serious adverse events), and AEs leading to discontinuation | Up to Day 8 of Period 3 (each period is 7 days; 3 periods total)
Number of Participants With Clinically Significant Change in Clinical Laboratory Values | Up to Day 8 of Period 3 (each period is 7 days; 3 periods total)
Number of Participants With Clinically Significant Change in Vital Signs | Up to Day 8 of Period 3 (each period is 7 days; 3 periods total)
Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) | Up to Day 8 of Period 3 (each period is 7 days; 3 periods total)
Number of Participants With Clinically Significant Change in Physical Examination | Up to Day 8 of Period 3 (each period is 7 days; 3 periods total)
Volume of distribution at terminal phase (VzF) of BMS-986278 and metabolite alone or in combination with pirfenidone | Up to Day 5 of period 3 (each period is 7 days; 3 periods total)
Time of maximum observed serum concentration (Tmax) of BMS-986278 and metabolite alone or in combination with pirfenidone | Up to Day 5 of period 3 (each period is 7 days; 3 periods total)
Elimination half-life (T-HALF) of BMS-986278 and metabolite alone or in combination with pirfenidone | Up to Day 5 of period 3 (each period is 7 days; 3 periods total)
Oral clearance (CL/F) of BMS-986278 and metabolite alone or in combination with pirfenidone | Up to Day 5 of period 3 (each period is 7 days; 3 periods total)
Time of maximum observed serum concentration (Tmax) of pirfenidone and metabolite alone or in combination with BMS-986278 | Up to Day 5 of Period 3 (each period is 7 days; 3 periods total)
Elimination half-life (T-HALF) of pirfenidone and metabolite alone or in combination with BMS-986278 | Up to Day 5 of Period 3 (each period is 7 days; 3 periods total)
Oral clearance (CL/F) of pirfenidone and metabolite alone or in combination with BMS-986278 | Up to Day 5 of Period 3 (each period is 7 days; 3 periods total)
Volume of distribution at terminal phase (VzF) Plasma Pharmokinetics of pirfenidone and metabolite alone or in combination with BMS-986278 | Up to Day 5 of Period 3 (each period is 7 days; 3 periods total)
Renal clearance (Clr) in Urine of pirfenidone alone or in combination with BMS-986278 | Up to Day 5 of Period 3 (each period is 7 days; 3 periods total)
Cumulative amount recovered in urine [Ae(0-T)] of pirfenidone alone or in combination with BMS-986278 | Up to Day 5 of Period 3 (each period is 7 days; 3 periods total)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences - Salt Lake, Salt Lake City, Utah, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm